CLINICAL TRIAL: NCT03866655
Title: Evaluating a Digital Tool for Supporting Breast Cancer Patients: A Prospective Randomised Controlled Trial
Brief Title: Evaluating a Digital Tool for Supporting Breast Cancer Patients
Acronym: ADAPT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Innovate UK (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CCR4965
Record Dates: First submitted 2019-02-19; First posted 2019-03-07 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Digital; eHealth; Supportive Care; Patient Activation; Resource Utilisation
MeSH Terms: conditions — Breast Neoplasms; Patient Participation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Device: OWise
- Control (No Intervention)

INTERVENTIONS:
Device: OWise — OWise Breast Cancer is a supportive care digital tool for breast cancer patients. The tool can be accessed as a mobile phone application or as a website. The tool has various tools for self-managing and self-monitoring treatment and symptoms such as an appointment calendar, a symptom-tracker, a modifiable question list and a recording device for consultations.
  Arms: Intervention

SUMMARY:
This is a prospective randomised controlled trial that aims to understand the impact of the OWise breast cancer digital tool in newly diagnosed breast cancer patients. Half the patients will receive the digital tool and half the patients will receive standard information. The study will look at the impact of the digital tool on patient activation, health related quality of life (HRQoL), health status, psychological distress, NHS resource utilisation and health care costs.

ELIGIBILITY:
Inclusion Criteria:

* female
* adult (age 18 years or over)
* newly diagnosed
* early breast cancer
* first primary cancer diagnosis
* under treatment at one of the participating sites.

Exclusion Criteria:

* have started anti-cancer treatment
* private patients
* unable to read or write in English
* significant cognitive impairment
* poor mental health
* do not have access to the internet
* confirmed metastatic disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Comparison of the change in patient activation (validated questionnaire: Patient Activation Measure (PAM-13) Survey) | 3 months after diagnosis (primary objective); 6 months and 1 year (secondary objective)
  The Patient Activation Measure (PAM-13) is a 13-item questionnaire measuring confidence in self management and knowledge of health condition. Each item has four possible responses from (1) strongly disagree to (4) strongly agree, with an additional 'not applicable' option. The measure views activation as a developmental process of four different levels, with the lowest scores corresponding to 'not believing activation important' and the highest scores corresponding to 'taking action.'
  The total score is calculated by dividing the raw score by the number of items answered (excluding items where 'not applicable' was selected) and multiplying by 13. This score is transformed using calibration tables to a scale with a theoretical range of 1-100, with a higher PAM score indicating higher patient activation.

SECONDARY OUTCOMES:
Comparison of the change in health status (validated questionnaire: EuroQol 5-Dimension 5-Level (EQ-5D-5L) Survey) | 3 months, 6 months and 1 year after diagnosis
  The EuroQol 5-Dimension 5-Level (EQ-5D-5L) questionnaire measures health status and includes the descriptive system and the EuroQol visual analogue scale (EQ VAS). The descriptive system has 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each has 5 levels of response resulting in a single digit number that expresses the level for that dimension (1-5): no problems, slight problems, moderate problems, severe problems and extreme problems. Combined, the digits for the 5 dimensions create a 5-digit number that describes the patient's health state. For each health state, a corresponding index value will be determined.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The worst health you can imagine' and 'The best health you can imagine' with numbers between 0 and 100. This score is a quantitative measure of health outcome that reflects the patient's own judgement.
Comparison of the change in health related quality of life (validated questionnaire: European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Core30 (EORTC-QLQ-C30 version 3) Survey) | 3 months, 6 months and 1 year after diagnosis
  The European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Core30 (EORTC-QLQ-C30 version 3) is a 30-item questionnaire measuring quality of life. It consists of five functional scales (physical, role, cognitive, emotional and social), a global quality of life scale, three symptom scales (fatigue, pain, nausea and vomiting), single items assessing common symptoms (dyspnea, loss of appetite, sleep disturbance, constipation and diarrhea) and a single item assessing perceived financial impact.
  After linear transformation, all scales and single item measures range in score from 0-100. A higher score on the functional scales and global quality of life scale indicates better function and HRQoL. A higher score on the symptom scales and items indicates higher symptom burden.
Comparison of the change in psychological distress (validated questionnaire: HADS) | 3 months, 6 months and 1 year after diagnosis
  The Hospital Anxiety and Distress Scale (HADS) questionnaire is a 14-item instrument measuring anxiety, depression and overall psychological distress, with seven items assessing anxiety and seven items assessing depression. Each item is scored from 0-3 and meaning a person can score between 0 and 21 for either anxiety or depression. The summed total score reflects the level of psychological distress. Higher total scores are indicative of more psychological distress.
  We will compare the mean change in each of the three scale scores in the intervention and control arm in simple and multiple linear regression models including potential covariates. Based on the continuous overall psychological distress score, patients are classified as 'distressed' when they have a score of ≥8, and 'not distressed' when they have a score <8.
Resource Utilisation | 1 year
  Number of primary, secondary and social care visits consumed by each patient. We will extract the total number of clinic or hospital visits to the general practitioner, secondary care, emergency departments, urgent care and social care. We will extract the average number of resources consumed by each patient and the average cost associated with each patient in total and stratified by commissioning group and secondary hospital.
  We will present the mean rate of resource utilisation in the two groups for the various types of resources (primary, secondary and social care) and for the total National Health Service (NHS) resources. The secondary analysis will compare the mean rate of total resource utilisation in the two groups in simple and multiple linear regression models including potential covariates.
Health care costs | 1 year
  Cost per patient according to clinical commissioning group. We will extract the average number of resources consumed by each patient and the average cost associated with each patient in total and stratified by commissioning group and secondary hospital.
  We will present the mean cost per patient in the two groups for the various types of resources (primary, secondary and social care) and for the total NHS resources. The secondary analysis will compare the mean cost per patient in the two groups in simple and multiple linear regression models including potential covariates.

CONTACTS AND LOCATIONS:
Overall Officials: Olga Husson, PhD, Principal Investigator — Institute of Cancer Research, United Kingdom
Locations (1):
- The Royal Marsden NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The patient reported outcomes will be available via the PROFILES Registry at the Royal Marsden NHS Foundation Trust.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will be available one year after study closure.
Access Criteria: The registry is accessible based on approval of specific research questions from the PROFILES Review and Management Group.

REFERENCES:
- [Derived] Vrancken Peeters NJMC, Georgopoulou S, Kulakowski R, Hainsworth E, Lidington E, McGrath SE, Noble J, Azarang L, Husson O, Cruickshank S. Effect of a digital tool on breast cancer specific health-related quality of life and psychological distress: secondary results from the ADAPT study. Support Care Cancer. 2025 Oct 8;33(11):916. doi: 10.1007/s00520-025-09968-8. PMID 41060446
- [Derived] Vrancken Peeters NJMC, Husson O, Kulakowski R, Hainsworth E, Lidington E, McGrath SE, Noble J, Azarang L, Cruickshank S, Georgopoulou S. Evaluating a digital tool for supporting people affected by breast cancer: a prospective randomized controlled trial-the ADAPT study. Support Care Cancer. 2024 Oct 21;32(11):740. doi: 10.1007/s00520-024-08923-3. PMID 39432189
- [Derived] Lidington E, McGrath SE, Noble J, Stanway S, Lucas A, Mohammed K, van der Graaf W, Husson O. Evaluating a digital tool for supporting breast cancer patients: a randomized controlled trial protocol (ADAPT). Trials. 2020 Jan 15;21(1):86. doi: 10.1186/s13063-019-3971-6. PMID 31941539